CLINICAL TRIAL: NCT06618898
Title: Orofacial Pain and Oral Health-related Quality of Life in Woodwind and Cello Musicians in German Orchestras
Brief Title: Orofacial Pain in Woodwind and Cello Musicians in German Orchestras
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Felix Marschner, Postdoctoral Researcher, University Medical Center Goettingen
Other Study IDs: 13/9/24
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Orofacial Pain; Sleep Problems
Keywords: Musicals; orchestra; orofacial pain; quality of life; stress; sleep disorders
MeSH Terms: conditions — Facial Pain; Parasomnias; Sleep Wake Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- oboe: Woodwind players in German professional orchestras who play the oboe
  Interventions: Other: online questionnaire
- flute: Woodwind players in German professional orchestras who play the flute
  Interventions: Other: online questionnaire
- clarinet: Woodwind players in German professional orchestras who play the clarinet
  Interventions: Other: online questionnaire
- bassoon: Woodwind players in German professional orchestras who play the bassoon
  Interventions: Other: online questionnaire
- cello: musicians in German professional orchestras who play the cello
  Interventions: Other: online questionnaire

INTERVENTIONS:
Other: online questionnaire — The online questionnaire includes demographic data: age, gender, instrument (oboe, flute, clarinet, bassoon, and cello), years of service, number of services in the last six months and specific questions about orofacial pain, sleep bruxism, stress experiences, and sleep quality.
  Other Names: questionnaire

SUMMARY:
Professional musicians in German professional orchestras represent a population group that has received little attention so far, despite being exposed to a variety of work-related factors that may pose potential health risks to the orofacial system. These factors include environmental noise, irregular working hours, tight schedules, and high demands for quality and discipline, all of which can lead to stress, sleep disturbances, and physical impairments. This prospective, non-interventional survey study aims to assess the health challenges faced by woodwind players (oboe, flute, clarinet, bassoon). It will explore the relationship between the type of instrument played, orofacial pain, sleep problems, and oral health-related quality of life (OHRQoL). Woodwind players, due to their playing techniques, may be more susceptible to orofacial complaints, which could negatively impact their quality of life. A control group of cellists, whose playing techniques put less strain on the orofacial system, will be used for comparison. Participation will be via an online questionnaire targeting musicians who have been employed in a German professional orchestra for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* musicians whose primary instruments are oboe, flute, clarinet, bassoon, or cello
* at least 12 months of employment or freelance work in the past 5 years with a German professional orchestra

Exclusion Criteria:

* consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional musicians whose primary instruments are oboe, flute, clarinet, bassoon, or cello in German professional orchestras.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Online-Questionnaire | 10 minutes
  Completion of a web based questionnaire; Oral health impact profile 14: minimum value 0 and maximum value 56, higher scores indicating poor oral health related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marschner F, Sokolowski A, Sokolowski A, Biermann J, Wiegand A. Orofacial pain and oral health-related quality of life in woodwind and cello musicians in German orchestras: an online based questionnaire study. J Occup Med Toxicol. 2025 Jun 6;20(1):19. doi: 10.1186/s12995-025-00467-4. PMID 40481603